CLINICAL TRIAL: NCT00597454
Title: An Access Delivery Model That Eliminates Barriers to Breast Cancer Care Delivery With Emphasis on the Coordination of Care Within and Between an Outpatient Screening Facility and a Diagnostic and Treatment Center
Brief Title: An Access Delivery Model That Eliminates Barriers to Breast Cancer Care Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Ralph Lauren Center for Cancer Care and Prevention (Other); North General Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 04-067
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Patient Navigation

INTERVENTIONS:
Other: Patient Navigation — we will conduct a detailed analysis of how the patient navigators' time is actually utilized by having them record a detailed log categorizing their activities as it relates to the elimination of recognized barriers to care. Second, we will measure the time interval from receipt of a suspicious mammogram to appropriate diagnostic evaluation and or treatment.
  We will measure the number of women who experience diagnostic and or treatment delay and whether the presence of a Patient Navigator enables delivery of coordinated care that avoids delays. Third, we will measure patients' satisfaction with aspects of their care, focusing particularly on care coordination using validated instruments designed for this purpose.

SUMMARY:
The purpose of the research is to examine the usefulness of using patient navigators in improving coordination of care between the Breast Examination Center in Harlem (BECH) and the Ralph Lauren Center for Cancer Care and Prevention (RLCCCP) for patients with a suspicious breast finding. This study will collect information to improve the role of the Patient Navigator, nonmedical staff that helps coordinate patient care. The study will also collect information to be used to help remove barriers that happen when several different institutions provide care.

DETAILED DESCRIPTION:
This purpose of this protocol is to systematically evaluate the role of Patient Navigators, non-medical personnel who assist in the coordination of care, for women attending a breast cancer screening clinic in Harlem who are found to have a suspicious result. The concept of patient navigation, developed by Dr. Harold Freeman, has been identified as a promising strategy to reduce disparities in health care for minorities and the underserved.

This protocol will evaluate the role of the Patient Navigator in coordinating care for women who are referred to the Ralph Lauren Center for Cancer Care and Prevention (RLCCCP) from the Breast Examination Center of Harlem (BECH). To achieve this, we propose four interrelated tasks. First, we will characterize in detail the specific nature of the activities of the Navigators as they remedy barriers to the receipt of breast cancer care. Secondly, we will determine whether the presence of the Navigator minimizes the percentage of patients with significant delays in receipt of necessary care. Third, we will measure patient satisfaction with care and their perceptions of the value of the Navigator. Finally, we will provide a baseline needs assessment of those (eligible) patients requiring pain and palliation services.

Specific Aims:

1. To characterize the role of Patient Navigators by defining the specific tasks and activities they perform in order to eliminate and/or reduce barriers to receipt of cancer care.
2. To evaluate how the presence of a Patient Navigator influences the time intervals from receipt of a suspicious screening mammogram or palpable breast mass to appropriate diagnosis and or treatment.
3. To measure patient's satisfaction with the coordination of care in the presence of a Patient Navigator.
4. To descriptively assess the pain and palliation needs of the population under study.

ELIGIBILITY:
Inclusion Criteria:

* Women with a suspicious screening finding
* Referred from Breast Examination Center of Harlem (BECH)

Exclusion Criteria:

* Women that were not initially seen at Breast Examination Center of Harlem (BECH)
* Women with normal breast screening findings

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Eval how Navigators spend time & specific tasks undertake to coordinate care.Specificatn of time intervals from receipt of suspicious screening mammogram to receipt of approp diagnostic eval.Pt satisfaction evaluatn take place w/in 1 month of i | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Harper, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center/Ralph Lauren Center for Cancer Care and Prevention
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org